CLINICAL TRIAL: NCT00123253
Title: A Phase 3 Multicenter, Double-Blind, Randomized, Placebo-Controlled Study Assessing the Efficacy and Safety of a 2 mg Dose of TH9507, a Growth Hormone Releasing Factor Analog, in HIV Patients With Excess of Abdominal Fat Accumulation
Brief Title: TH9507 in Patients With HIV-Associated Lipodystrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Theratechnologies (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TH9507/III/LIPO/010; NCT00435136 (obsolete NCT alias)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: HIV; Lipodystrophy; Abdominal fat accumulation; Growth hormone releasing factor/Growth hormone releasing hormone; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — tesamorelin

INTERVENTIONS:
Drug: TH9507

SUMMARY:
HIV lipodystrophy affects a significant proportion of patients treated with combination antiretroviral therapy (ART) and is characterized by excess visceral fat accumulation and loss of extremity and subcutaneous fat, in association with dyslipidemia and insulin resistance. Data from a previous randomized, placebo-controlled trial demonstrated that daily administration of 2mg TH9507, a growth hormone releasing factor (GRF), to HIV patients with an excess of abdominal fat accumulation for 12 weeks resulted in decreases in visceral adipose tissue (VAT) and trunk fat, with no significant changes in limb fat and subcutaneous adipose tissue (SAT). This study is aimed at further assessing the efficacy and safety of 2 mg TH9507 in a larger population of HIV patients treated with ART and experiencing an excess of abdominal fat accumulation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 65 years inclusive
* HIV positive; CD4 cell counts >100 cells/mm3; viral load <10,000 copies/mL (stable for 8 weeks)
* On stable ART regimen for at least 8 weeks prior to randomization
* Have evidence of abdominal fat accumulation defined by the following anthropometric cut off values:

  * For males: waist circumference > 95 cm and waist to hip ratio > 0.94;
  * For females: waist circumference > 94 cm and waist to hip ratio > 0.88.
* Females of childbearing potential not pregnant or lactating; normal mammography within 6 months of study.
* Signed informed consent

Exclusion Criteria:

* Body mass index < 20 kg/m2
* Opportunistic infection; HIV-related disease within 3 months of study.
* History of malignancy; active neoplasm.
* Prostate-specific antigen (PSA) >5 ng/mL at screening
* Hypopituitarism; history of pituitary tumor/surgery; head irradiation; head trauma that has affected the somatotropic axis.
* Untreated hypothyroidism
* Type 1 diabetics and type 2 diabetics on oral hypoglycemic or insulin sensitizing agent within 6 months of study
* ALT or AST > 3 x ULN; serum creatinine > 133 mmol/L (1.5 mg/dL); hemoglobin more than 20 g/L below LLN; fasting blood glucose > 8.33 mmol/L (150 mg/dL); fasting triglycerides > 11.3 mmol/L (0.99 g/dL).
* Untreated hypertension
* Change in anti-hyperlipemic regimen within 3 months prior to study
* Change in testosterone regimen and/or supraphysiological dose of testosterone
* Estrogen therapy
* Anoretics/anorexigenics or anti-obesity agents within 3 months of study
* Growth hormone (GH); GH secretagogues; growth hormone releasing factor (GRF) products; IGF-1; or IGFBP-3 within 6 months of study.
* Drug or alcohol dependence or use of methadone within 6 months of study entry
* Participation in a clinical trial with any investigational drug/device within 30 days of screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2005-06; Primary Completion 2006-11 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Visceral adipose tissue (VAT)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (42):
- United States (35):
  - UCLA School of Medicine, Los Angeles, California
  - Office of Dr. Michael Somero, Palm Springs, California
  - UCSD Medical Center, San Diego, California
  - Kaiser Permanente, San Francisco, California
  - AIDS Research Alliance, West Hollywood, California
  - Capital Medical Associates, Washington D.C., District of Columbia
  - Bach & Godofsky, Bradenton, Florida
  - Office of Dr. Gary Richmond, Fort Lauderdale, Florida
  - Care Resource Miami, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infectious Disease Associates, Sarasota, Florida
  - Treasure Coast Infectious Disease Consultant (TDIDC), Vero Beach, Florida
  - AIDS Research Consortium Atlanta (ARCA), Atlanta, Georgia
  - Northern Healthcare, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Department of Medicine, Indianapolis, Indiana
  - Institute of Human Virology, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Community Research Initiative of New England, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Tufts University School of Medicine, Boston, Massachusetts
  - Community Research Initiative of New England (CRI West), Springfield, Massachusetts
  - Hennepin County Medical Centre, Minneapolis, Minnesota
  - AIDS Community Research Initiative of America, New York, New York
  - Bellevue Hospital Center New York University, New York, New York
  - St Luke's Roosevelt Hospital Centre, New York, New York
  - St Vincent Catholic Medical Centre, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Fanno Creek Clinic, LLC, Portland, Oregon
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - Dallas VA Medical Centre, Dallas, Texas
  - The University of Texas Medical School, Houston, Texas
  - Infectious Disease Physicians Inc., Annandale, Virginia
  - Swedish Medical Center, Seattle, Washington
- Canada (7):
  - Southern Alberta Clinic, Calgary, Alberta
  - St-Paul's Hospital, Vancouver, British Columbia
  - Sunnybrook and Women College Health Sciences Centre, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Clinique Médicale du Quartier Latin, Montreal, Quebec
  - Clinique Médicale L'Actuel, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Fourman LT, Czerwonka N, Feldpausch MN, Weiss J, Mamputu JC, Falutz J, Morin J, Marsolais C, Stanley TL, Grinspoon SK. Visceral fat reduction with tesamorelin is associated with improved liver enzymes in HIV. AIDS. 2017 Oct 23;31(16):2253-2259. doi: 10.1097/QAD.0000000000001614. PMID 28832410
- [Derived] Stanley TL, Falutz J, Marsolais C, Morin J, Soulban G, Mamputu JC, Assaad H, Turner R, Grinspoon SK. Reduction in visceral adiposity is associated with an improved metabolic profile in HIV-infected patients receiving tesamorelin. Clin Infect Dis. 2012 Jun;54(11):1642-51. doi: 10.1093/cid/cis251. Epub 2012 Apr 10. PMID 22495074
- [Derived] Falutz J, Mamputu JC, Potvin D, Moyle G, Soulban G, Loughrey H, Marsolais C, Turner R, Grinspoon S. Effects of tesamorelin (TH9507), a growth hormone-releasing factor analog, in human immunodeficiency virus-infected patients with excess abdominal fat: a pooled analysis of two multicenter, double-blind placebo-controlled phase 3 trials with safety extension data. J Clin Endocrinol Metab. 2010 Sep;95(9):4291-304. doi: 10.1210/jc.2010-0490. Epub 2010 Jun 16. PMID 20554713
- [Derived] Falutz J, Potvin D, Mamputu JC, Assaad H, Zoltowska M, Michaud SE, Berger D, Somero M, Moyle G, Brown S, Martorell C, Turner R, Grinspoon S. Effects of tesamorelin, a growth hormone-releasing factor, in HIV-infected patients with abdominal fat accumulation: a randomized placebo-controlled trial with a safety extension. J Acquir Immune Defic Syndr. 2010 Mar;53(3):311-22. doi: 10.1097/QAI.0b013e3181cbdaff. PMID 20101189
- [Derived] Falutz J, Allas S, Blot K, Potvin D, Kotler D, Somero M, Berger D, Brown S, Richmond G, Fessel J, Turner R, Grinspoon S. Metabolic effects of a growth hormone-releasing factor in patients with HIV. N Engl J Med. 2007 Dec 6;357(23):2359-70. doi: 10.1056/NEJMoa072375. PMID 18057338